CLINICAL TRIAL: NCT01203748
Title: Substrate and Trigger Ablation for Reduction of Atrial Fibrillation Trial - Star AF II Study
Acronym: Star AF II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AF-09-102-ID-AB
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PVI + Lines Ablation (Experimental)
  Interventions: Procedure: PVI + Lines ablation
- PVI Ablation (Active Comparator)
  Interventions: Procedure: PVI
- PVI + CFE (Experimental)
  Interventions: Procedure: PVI + CFE ablation

INTERVENTIONS:
Procedure: PVI + Lines ablation — Pulmonary vein antrum isolation with additional linear ablation (mitral line and roof line)
  Arms: PVI + Lines Ablation
Procedure: PVI — Pulmonary vein antrum isolation
  Arms: PVI Ablation
Procedure: PVI + CFE ablation — Pulmonary vein antrum isolation with additional complex fractionated electrogram ablation
  Arms: PVI + CFE

SUMMARY:
This investigation is designed with the hypothesis that combined PV Antral Isolation and Ablation of Complex Fractionated Electrograms (PVI+CFE) approach will offer a higher success rate compared to the Wide Circumferential Pulmonary Vein Antrum Isolation (PVI) approach and to the Combined PV Antral Isolation and Empiric Linear Ablation (PVI+Lines) approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients age is18 years or greater;
* Patients undergoing a first-time ablation procedure for AF;
* Patients with persistent AF;
* Persistent AF will be defined as a sustained episode lasting > 7 days and less than 3 years.
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication;
* At least one episode of persistent AF must have been documented by ECG, holter, loop recorder, telemetry, trans telephonic monitoring (TTM), or implantable device within last 2 years of enrollment in this investigation;
* Patients must be able and willing to provide written informed consent to participate in this investigation; and
* Patients must be willing and able to comply with all peri-ablation and follow-up requirements.

Exclusion Criteria:

* Patients with paroxysmal AF;
* Patients with long-standing persistent AF;
* Patients for whom cardioversion or sinus rhythm will never be attempted/pursued;
* Patients with AF felt to be secondary to an obvious reversible cause;
* Patients with contraindications to systemic anticoagulation with heparin or coumadin or a direct thrombin inhibitor;
* Patients with left atrial size ≥ 60 mm (2D echocardiography, parasternal long axis view); and
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Freedom from AF | 18 months
  Freedom from documented AF episodes > 30 seconds at 18 months after one or two ablation procedure with/without antiarrhythmic medications (AAD).
  In the CT.gov website and in our protocol, we have stated the above primary endpoint (PE). This was the identical PE used in the original STAR AF I study. The intent of this PE was to present the success rates after both 1 procedure and after 2 procedures separately as was done in the original STAR AF I study. However, this is not entirely clear from the way the PE is stated. It may appear that our PE is the success rate after 2 procedures ("1 or 2" may imply "2"). Since our sample size calculation for the STAR AF II study was based on a single procedure success rate, the single procedure success rate with/without AAD will be used as the PE. The success rate after 2 procedures will be provided as the 1st. secondary endpoint. This clarification is done prior to locking the database and prior to any data analysis.

SECONDARY OUTCOMES:
Freedom from atrial arrhythmia | 18 months
  Freedom from documented atrial arrhythmia episodes > 30 seconds at 18 months after one or two ablation procedures with/without antiarrhythmic medications
Freedom from atrial flutter and AT | 18 months
  Freedom from documented atrial flutter and atrial tachycardia episodes > 30 seconds at 18 months after one and two procedures with/without antiarrhythmic medications
Freedom from documented or not atrial arrhythmia | 18 months
  Freedom from any atrial arrhythmia (documented or not) episodes > 30 seconds at 18 months after one or two ablation procedures with/without antiarrhythmic medications
Freedom from symptomatic AF | 18 months
  Freedom from symptomatic AF episodes > 30 seconds at 18 months after one or two ablation procedures with/without antiarrhythmic medications
Freedom from symptomatic atrial arrhythmia | 18 months
  Freedom from symptomatic atrial arrhythmia episodes > 30 seconds at 18 months after one or two ablation procedures with/without antiarrhythmic medications
Incidence of peri-procedural complications, including stroke, PV stenosis, cardiac perforation, esophageal injury and death | 18 months
  Incidence of peri-procedural complications, including stroke, PV stenosis, cardiac perforation, esophageal injury and death
Procedure duration and fluoroscopy time | 18 months
  Procedure duration and fluoroscopy time
Number of repeat procedures | 18 months
  Number of repeat procedures
Effect of each strategy on AF cycle length/regularity/termination | 18 months
  Effect of each strategy on AF cycle length/regularity/termination
Relationship of acute termination of AF to long-term procedural outcome | 18 months
  Relationship of acute termination of AF to long-term procedural outcome
Percentage achievement of complete linear block in linear ablation arm | 18 months
  Percentage achievement of complete linear block in linear ablation arm
Effect of complete linear block on procedural outcome in linear ablation arm | 18 months
  Effect of complete linear block on procedural outcome in linear ablation arm
Quality of life measurements (SF-36, EQ-5D and CCS SAF) | 18 MONTHS
  Quality of life measurements (SF-36, EQ-5D and CCS SAF) at baseline, 6, 12 and 18 months after one and/or two ablation procedures
Correlation of AF burden to symptoms and quality of life changes | 18 Months
  Correlation of AF burden to symptoms and quality of life changes
Improvement in AF burden by > 90% post ablation procedure | 18 months
  Improvement in AF burden by > 90% post ablation procedure
Relationship of ablating all atrial arrhythmias versus ablation of only targeted endpoints on long term outcome | 18 months
  Relationship of ablating all atrial arrhythmias versus ablation of only targeted endpoints on long term outcome
Cut off of AF burden that affects the Quality of Life measurement | 18 months
  Cut off of AF burden that affects the Quality of Life measurement
Evaluation of cost utility | 18 months
  Evaluation of cost utility

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, Dr., Principal Investigator — Southlake Regional Health Centre
Locations (2):
- St. Andrews War Memorial Hospital, Brisbane, Queensland, Australia
- Southlake Regional Health Centre, Newmarket, Ontario, Canada

REFERENCES:
- [Derived] Terricabras M, Mantovan R, Jiang CY, Betts TR, Chen J, Deisenhofer I, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P, Verma A; Substrate and Trigger Ablation for Reduction of Atrial Fibrillation Trial-Part II (STAR AF II) Investigators. Association Between Quality of Life and Procedural Outcome After Catheter Ablation for Atrial Fibrillation: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2025473. doi: 10.1001/jamanetworkopen.2020.25473. PMID 33275151
- [Derived] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Derived] Verma A, Sanders P, Macle L, Deisenhofer I, Morillo CA, Chen J, Jiang CY, Ernst S, Mantovan R. Substrate and Trigger Ablation for Reduction of Atrial Fibrillation Trial-Part II (STAR AF II): design and rationale. Am Heart J. 2012 Jul;164(1):1-6.e6. doi: 10.1016/j.ahj.2012.04.002. PMID 22795275